CLINICAL TRIAL: NCT04253262
Title: A Phase Ib/II Study of Copanlisib Combined With Rucaparib in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Copanlisib Combined With Rucaparib in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Bayer (Industry); Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 360
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — rucaparib; copanlisib

STUDY DESIGN:
Intervention Model Description: Dose escalation will follow the standard 3+3 design. Once the maximum tolerated dose is achieved in Phase I, Phase II will proceed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose Level -2 (Experimental): 300 mg Rucaparib, 45 mg (day 1 & 15) Copanlisib
  Interventions: Drug: Rucaparib; Drug: Copanlisib
- Dose Level -1 (Experimental): 400 mg Rucaparib, 45 mg (day 1 & 15) Copanlisib
  Interventions: Drug: Rucaparib; Drug: Copanlisib
- Dose Level 1 (Experimental): 400 mg Rucaparib, 45 mg Copanlisib
  Interventions: Drug: Rucaparib; Drug: Copanlisib
- Dose Level 2 (Experimental): 500 mg Rucaparib, 45 mg Copanlisib
  Interventions: Drug: Rucaparib; Drug: Copanlisib
- Dose Level 3 (Experimental): 600 mg Rucaparib, 45 mg Copanlisib
  Interventions: Drug: Rucaparib; Drug: Copanlisib
- Dose Level 4 (Experimental): 600 mg Rucaparib, 60 mg Copanlisib
  Interventions: Drug: Rucaparib; Drug: Copanlisib

INTERVENTIONS:
Drug: Rucaparib — Rucaparib (PO twice daily continuous)
  Other Names: Rubraca
Drug: Copanlisib — Copanlisib (IV day 1, 8, 15; 28 day cycle)
  Other Names: Aliqopa

SUMMARY:
This is a single arm Phase Ib/II, open label, safety, pharmacokinetic and efficacy clinical study in adult patients with metastatic castration-resistant prostate cancer (mCRPC). Patients will be treated with the combination of copanlisib and rucaparib for as long as the patient does not have clinically significant progressive disease and/or unacceptable toxicity and/or as long as the investigator deems that the patient is benefiting from treatment. Treatment may also be stopped if the patient withdraws consent, or study termination occurs.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
3. Life expectancy of at least 3 months
4. Histologically confirmed prostate cancer. Treatment-emergent small cell/NEPC (neuroendocrine prostate cancer) is allowed, but de novo small cell carcinoma of the prostate is excluded.
5. Progressive metastatic prostate cancer despite castrate levels of testosterone (< 50 ng/dL).
6. Patients may have either non-measurable disease OR measurable disease (by RECIST criteria)
7. Progressive disease during treatment (or within 4 weeks of completion) with abiraterone, enzalutamide, and/or apalutamide based on any one of the following:

   * For patients with measurable disease, progression by the RECIST 1.1 criteria
   * PSA evidence for progressive prostate cancer consists of a PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least one week apart. If the confirmatory PSA value is less than the screening PSA value, then an additional test for rising PSA will be required to document progression for the purposes of eligibility
   * Radionuclide bone scan: At least two new foci consistent with metastatic lesions
8. Testosterone < 50 ng/dL. Patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone bilateral orchiectomy.
9. Prior therapy with taxane in the castrate-sensitive or castration-resistant settings will be allowed. Prior treatment with radium-223 or sipuleucel-T is permitted, but not required.
10. No other systemic therapies for prostate cancer within 21 days prior to cycle 1 day 1 of study therapy or 5 half-lives, whichever is shorter, prior to day 1 of study therapy.
11. Left ventricular ejection fraction (LVEF) ≥ 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) obtained during screening
12. Patients must have adequate organ and bone marrow function within 14 days of inclusion in the study as defined below:

    * Absolute Neutrophil Count ≥ 1,500/mm3
    * Hemoglobin ≥ 9 g/dL
    * Platelets ≥ 100,000 /mm3
    * PT/INR ≤ 1.5 x ULN unless on chronic and stable anticoagulation at time of study entry
    * Bilirubin ≤1.5 x institutional upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's Syndrome, who can have total bilirubin <3.0 mg/dL
    * AST/ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases present)
    * Lipase ≤ 1.5 x ULN
    * HbA1c < 8.5 %
    * Serum Creatinine ≤ 1.5 X ULN (upper limit of normal) or creatinine clearance ≥ 45 mL/minute (using Cockcroft/Gault formula)
13. Sexually active males must use a condom with spermicide during intercourse while taking the drug and for 6 months after stopping treatment, even if patient is vasectomized to prevent delivery of the drug via seminal fluid.
14. Patients must agree to provide tumor tissue, either fresh or archival specimen of primary tumor and/or metastatic lesion, if available. Availability of tissue will not be required for enrollment.
15. Subjects must have the ability to understand and the willingness to sign a written informed consent prior to registration on study. Subjects should be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations at the institution.
16. Only during phase 2, patients will be required to have mutations in DNA repair genes based on molecular tests performed on germline DNA, prostate cancer tissue or ctDNA. Qualifying mutations (i.e. deleterious/pathogenic alterations) in at least one of the following genes involved with homologous recombination repair will be required: BRCA1, BRCA2, ATM, BARD1, BRIP1, CDK12, CHEK1, FANCL, FANCA, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, and RAD54L. Variants of unknown significance in one of the above genes are not eligible.

Exclusion Criteria

1. History of myelodysplastic syndrome or acute myeloid leukemia.
2. During phase 2, patients must not have received previous treatment with a DNA-damaging cytotoxic chemotherapy (e.g. prior platinum-based chemotherapy and mitoxantrone are not permitted) or PARP inhibitor. Prior treatment with PARP inhibitor is allowed during phase I dose escalation.
3. Untreated leptomeningeal or metastatic CNS disease; patients with treated disease may be eligible if clinically stable for 4 weeks after radiation or surgery including those with history of spinal cord compression that have received definitive treatment. If patients are receiving steroids as adjunct for treatment of leptomeningeal disease or metastatic CNS disease, dose should be stable for 4 weeks prior to day 1 of cycle 1.
4. Clinically significant, uncontrolled heart disease and/or recent events including any of the following:

   * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 6 months prior to screening
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening. Patients with rate-controlled atrial fibrillation or flutter are permitted.
   * QTcF > 470 msec on screening 12-lead ECG
   * Documented cardiomyopathy
5. Clinically significant uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management). For the purpose of this protocol definition of uncontrolled hypertension is based on persistent (≥72 hours) and symptomatic.
6. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication. However, patients with a venous thrombosis, including a pulmonary embolus, who have been on stable anticoagulation (more than 1 month without bleeding on a stable dose) is permitted. Patients with evidence or history of uncontrolled bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication
7. History or concurrent condition of clinically significant interstitial lung disease and/or severely impaired lung function. History of renal failure requiring peritoneal dialysis or hemodialysis. History of cirrhosis Child-Pugh B or C. Intestinal malabsorption.
8. Active, clinically serious infections of CTCAE (v 5.0) Grade ≥ 2 or per investigator discretion.
9. History of uncontrolled human immunodeficiency virus (HIV) infection defined as CD4 < 200 cells/mm3 or detectable viral load is not allowed.
10. Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel. Patients positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA. These patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.
11. Previous or concurrent history of malignancies within 5 years prior to study treatment except for curatively treated cervical carcinoma in situ, non-melanoma skin cancer, superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria]) or other T1 tumor that has been surgically removed with a low chance of recurrence in the next 3 years.
12. Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation
13. Ongoing substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
14. Prior radiation within 7 days of start drug. Prior major surgery, open biopsy or significant trauma within 28 days of start drug.
15. Patients with severe psychiatric illness/social situations that would limit compliance with study requirements in the judgment of study investigator
16. Patient has a history of non-compliance to medical regimen or inability to grant consent
17. Ongoing immunosuppressive therapy. Patients may be receiving up to 10mg/day of prednisone.
18. Radiotherapy or immuno-/chemotherapy less than 2 weeks before start of treatment. A wash-out period of 2 months from radiopharmaceuticals such as radium-223 and 177Lu-PSMA among others will be required.
19. Myeloid growth factors within 14 days prior to treatment.
20. Blood or platelet transfusion less than 7 days before cycle 1 day 1.
21. History of having received an allogeneic bone marrow or organ transplant.
22. Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of treatment, or have not recovered from major side effects; open biopsy within 7 days before start of treatment.
23. Anti-arrhythmic therapy for ventricular arrhythmias. Use of amiodarone and propafenone for atrial fibrillation rate control is allowed.
24. Use of CYP3A4 inhibitors and inducers. Copanlisib is primarily metabolized by CYP3A4. Therefore concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, darunavir, indinavir, lopinavir, mifepristone, posaconazole, ombitasvir, idelalisib, cobicistat, atazanavir, ritonavir, indinavir, nelfinavir and saquinavir) and inducers (apalutamide, carbamazepine, enzalutamide, fosphenytoin, phenobarbital, phenytoin, primidone, rifampin) is not allowed. Rucaparib is a moderate inhibitor of CYP1A2 and a weak inhibitor of CYP2C9, CYP2C19 and CYP3A4 and no specific medications is contra-indicated but dose adjustment may be necessary of concurrent medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Cycle 1 (each cycle is 28 days) through pre-dosing cycle 2, approximately 1 month.
  To evaluate the maximum tolerated dose of copanlisib with rucaparib in patients with metastatic castration-resistant prostate cancer.
Response | Every 28 days on treatment, then every 3 months until progression of disease up to 3 years.
  To estimate the overall response rate of the combination of copanlisib and rucaparib in patients with metastatic castration-resistant prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Benedito Carneiro, MD, MS, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Helen Diller Family Comprehensive Cancer Center University of California San Francisco, San Francisco, California
  - Lifespan Cancer Institute, Providence, Rhode Island